CLINICAL TRIAL: NCT00519220
Title: Short and Long Term Outcomes of Heller Myotomy
Brief Title: Outcome of Symptoms in Patients Undergoing a Heller Myotomy
Acronym: Achalasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kenneth Luberice, Principal Investigator, University of South Florida
Other Study IDs: 105235
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Achalasia
Keywords: achalasia, Heller myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: Patients will answer symptom questionnaires and have their charts reviewed for relevant medical information.
  Interventions: Other: Symptom questionnaire

INTERVENTIONS:
Other: Symptom questionnaire — Patients will answer questionnaires evaluating their symptoms of achalasia.

SUMMARY:
The objective of this study is to review studies and patient symptoms before and after laparoscopic Heller myotomy to assess outcomes following laparoscopic surgery for achalasia.

DETAILED DESCRIPTION:
Patients will answer questionnaires before and after surgery to evaluate their symptoms of achalasia and will also have their charts reviewed for relevant medical information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with achalasia who have had laparoscopic Heller myotomies for the treatment of achalasia

Exclusion Criteria:

* No patients under the age of 18 will be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with achalasia who have had laparoscopic Heller myotomies at Tampa General Hospital.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2006-12; Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The objective of this study is to review pre-operative and post-operative studies and patient evaluation reports to evaluate patient outcomes following laparoscopic surgery for achalasia | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Rosemurgy, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital/University of South Florida, Tampa, Florida, United States